CLINICAL TRIAL: NCT05913427
Title: Prospective, Phase II Study to Evaluate the Efficacy of Addition of Progesterone to Standard Chemotherapy According to Etoposide-Doxorubicin-Cisplatin Scheme Plus Mitotane (EDP-M) in Patients With Advanced Adrenocortical Carcinoma (ACC)
Brief Title: Evaluation of the Efficacy of Addition of Progesterone to Standard Chemotherapy in Adrenocortical Carcinoma (ACC)
Acronym: PESETA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Principal Investigator, Alfredo Berruti, Medical Oncologist, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ASSTBS-FARONCO- PESETA-20
Record Dates: First submitted 2023-03-07; First posted 2023-06-22 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Adrenocortical Carcinoma
MeSH Terms: conditions — Adrenocortical Carcinoma | interventions — Etoposide; Doxorubicin; Cisplatin; Mitotane; Megestrol Acetate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EDP-M plus MEGESTROL ACETATE 160 mg (Experimental): EDP will be administered at the following doses: doxorubicin 40 mg/m2 on day 1, etoposide 100 mg/m2 days 2-4, cisplatin 40 mg/m2 days 3-4, every 28 days. Concomitant mitotane therapy will be administered continuously. Megestrole 160 mg 2 tablets will be administered once daily (in the morning) and will be stopped 21 days after the last administration of the EDP.
  Interventions: Drug: Etoposide, doxorubicin, cisplatin and Mitotane plus Megestrol Acetate 160 MG
- EDP-M plus PLACEBO (Placebo Comparator): EDP will be administered at the following doses: doxorubicin 40 mg/m2 on day 1, etoposide 100 mg/m2 days 2-4, cisplatin 40 mg/m2 days 3-4, every 28 days. Concomitant mitotane therapy will be administered continuously. Placebo 2 tablets will be administered once daily (in the morning) and will be stopped 21 days after the last administration of the EDP.
  Interventions: Drug: Etoposide, doxorubicin, cisplatin and Mitotane plus Placebo

INTERVENTIONS:
Drug: Etoposide, doxorubicin, cisplatin and Mitotane plus Megestrol Acetate 160 MG — EDP will be administered at the following doses: doxorubicin 40 mg/m2 on day 1, etoposide 100 mg/m2 days 2-4, cisplatin 40 mg/m2 days 3-4, every 28 days.
  Megestrol acetate will be prepared and packaged by the authorized external contract development and manufacturing organization (CDMO) Doppel Farmaceutici s.r.l. (Cortemaggiore, PC), that, according to the GMP and applicable law (FU XII ed) will also prepare the related placebo, in accordance with GMP (annex 13) and applicable law (FU XII ed.).
  Other Names: Megace
  Arms: EDP-M plus MEGESTROL ACETATE 160 mg
Drug: Etoposide, doxorubicin, cisplatin and Mitotane plus Placebo — EDP will be administered at the following doses: doxorubicin 40 mg/m2 on day 1, etoposide 100 mg/m2 days 2-4, cisplatin 40 mg/m2 days 3-4, every 28 days. Placebo 160 mg tablets will be developed by the CDMO to have the same appearance and taste as the tablet containing the active drug.
  Other Names: placebo
  Arms: EDP-M plus PLACEBO

SUMMARY:
This is a prospective randomized, double blind, placebo controlled phase II study planned in patients with advanced ACC. The study will be conducted at ASST Spedali Civili Hospital and University of Brescia in Brescia.

DETAILED DESCRIPTION:
As no effective second-line therapies are available for patients with disease progression to EDPM, including modern molecular target therapies and immunotherapy, it is reasonable to expect that no newer drugs or combination regimens will be able to replace EDPM in the next 5 years. Since EDP-M is destined to remain the standard first line therapy, research strategies aimed to improve the efficacy of this regimen are of relevance. In this study, investigators will address the hypotheses that progesterone has a synergistic and/or additive effect to EDP-M in inducing cytotoxicity in ACC cells in vitro and the antineoplastic activity of EDP-M in locally advanced/metastatic ACC patients could be improved by the addition of megestrol acetate.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of ACC
* Locally advanced or metastatic disease not amenable to radical surgery resection
* ECOG performance status 0-2
* Effective contraception
* Life expectancy > 3 months
* Age > 18 years
* Adequate bone marrow reserve (neutrophils >1,000/mm3 and/or platelets >80,000/mm3) and organ function (including renal, liver and cardiac function)
* Be able to comply with the protocol procedures and provide written informed consent.

Exclusion Criteria:

* History of recent or active prior malignancy, except for cured non-melanoma skin cancer, cured in situ cervical carcinoma, breast ductal carcinoma in situ, or other treated malignancies where there has been no evidence of disease for at least 2 years
* Renal insufficiency (estimated glomerular filtration rate [GFR]<50 mL/min/1.73 m2) or significant liver insufficiency (serum bilirubin>2 times the upper normal range and/or serum alanine aminotransferase [ALT] or aspartate aminotransferase [AST]>3 times the upper normal range). GFRs will be calculated according to the validated formula (MDRD)
* Pregnancy or breast feeding
* Congestive heart failure (ejection fraction<45%)
* Preexisting grade 2 peripheral neuropathy
* Previous or current treatment with mitotane or other antineoplastic drugs for ACC
* Previous radiotherapy for ACC
* Any other severe acute or chronic medical or psychiatric condition or laboratory abnormality that would impart, in the judgment of the investigator, excess risk associated with study participation or study drug administration or that, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-06-08 (Actual); Primary Completion 2027-06-08 (Estimated); Study Completion 2027-06-08 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the activity of the combination regimen (EDP-M plus progesterone (EDP-MP) versus EDP-M plus placebo) in advanced/ metastatic patients with ACC. | 18 months
  Comparison of proportion of patients attaining an Objective Response (Objective Response Rate, ORR), evaluated by RECIST criteria between the 2 treatment arms.

SECONDARY OUTCOMES:
Evaluation of the impact of the combination of the two treatments on hormone response in patients with secreting ACC; | 18 months
  Changes in serum cortisol from baseline in the two treatment arms;
Evaluation of the impact of the combination of the two treatments on hormone response in patients with secreting ACC; | 18 months
  Changes in serum UFC from baseline in the two treatment arms;
Evaluation of the impact of the combination of the two treatments on hormone response in patients with secreting ACC; | 18 months
  Changes in serum salivary cortisol from baseline in the two treatment arms;
Evaluation of the impact of the combination of the two treatments on hormone response in patients with secreting ACC; | 18 months
  Changes in ACTH from baseline in the two treatment arms;
Evaluation of the impact of the combination of the two treatments on hormone response in patients with secreting ACC; | 18 months
  Changes in serum 11-deoxycortisol from baseline in the two treatment arms;
Evaluation of the impact of the combination of the two treatments on hormone response in patients with secreting ACC; | 18 months
  Changes in serum aldosterone from baseline in the two treatment arms;
Evaluation of the impact of the combination of the two treatments on hormone response in patients with secreting ACC; | 18 months
  Changes in serum PRA from baseline in the two treatment arms;
Evaluation of the impact of the combination of the two treatments on hormone response in patients with secreting ACC; | 18 months
  Changes in serum androstenedione from baseline in the two treatment arms;
Evaluation of the impact of the combination of the two treatments on hormone response in patients with secreting ACC; | 18 months
  Changes in serum DHEA-S from baseline in the two treatment arms;
Evaluation of the impact of the combination of the two treatments on hormone response in patients with secreting ACC; | 18 months
  Changes in serum progesterone from baseline in the two treatment arms;
Evaluation of the impact of the combination of the two treatments on hormone response in patients with secreting ACC; | 18 months
  Changes in serum total testosterone from baseline in the two treatment arms;

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Berruti, Principal Investigator — ASST Spedali Civili di Brescia
Locations (1):
- Alfredo Berruti, Brescia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fassnacht M, Assie G, Baudin E, Eisenhofer G, de la Fouchardiere C, Haak HR, de Krijger R, Porpiglia F, Terzolo M, Berruti A; ESMO Guidelines Committee. Electronic address: clinicalguidelines@esmo.org. Adrenocortical carcinomas and malignant phaeochromocytomas: ESMO-EURACAN Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2020 Nov;31(11):1476-1490. doi: 10.1016/j.annonc.2020.08.2099. Epub 2020 Aug 27. No abstract available. PMID 32861807
- [Result] Fassnacht M, Terzolo M, Allolio B, Baudin E, Haak H, Berruti A, Welin S, Schade-Brittinger C, Lacroix A, Jarzab B, Sorbye H, Torpy DJ, Stepan V, Schteingart DE, Arlt W, Kroiss M, Leboulleux S, Sperone P, Sundin A, Hermsen I, Hahner S, Willenberg HS, Tabarin A, Quinkler M, de la Fouchardiere C, Schlumberger M, Mantero F, Weismann D, Beuschlein F, Gelderblom H, Wilmink H, Sender M, Edgerly M, Kenn W, Fojo T, Muller HH, Skogseid B; FIRM-ACT Study Group. Combination chemotherapy in advanced adrenocortical carcinoma. N Engl J Med. 2012 Jun 7;366(23):2189-97. doi: 10.1056/NEJMoa1200966. Epub 2012 May 2. PMID 22551107
- [Result] Fiorentini C, Fragni M, Perego P, Vezzoli S, Bonini SA, Tortoreto M, Galli D, Claps M, Tiberio GA, Terzolo M, Missale C, Memo M, Procopio G, Zaffaroni N, Berruti A, Sigala S. Antisecretive and Antitumor Activity of Abiraterone Acetate in Human Adrenocortical Cancer: A Preclinical Study. J Clin Endocrinol Metab. 2016 Dec;101(12):4594-4602. doi: 10.1210/jc.2016-2414. Epub 2016 Sep 14. PMID 27626976
- [Result] Fragni M, Fiorentini C, Rossini E, Fisogni S, Vezzoli S, Bonini SA, Dalmiglio C, Grisanti S, Tiberio GAM, Claps M, Cosentini D, Salvi V, Bosisio D, Terzolo M, Missale C, Facchetti F, Memo M, Berruti A, Sigala S. In vitro antitumor activity of progesterone in human adrenocortical carcinoma. Endocrine. 2019 Mar;63(3):592-601. doi: 10.1007/s12020-018-1795-x. Epub 2018 Oct 26. PMID 30367443
- [Result] Rossini E, Tamburello M, Abate A, Beretta S, Fragni M, Cominelli M, Cosentini D, Hantel C, Bono F, Grisanti S, Poliani PL, Tiberio GAM, Memo M, Sigala S, Berruti A. Cytotoxic Effect of Progesterone, Tamoxifen and Their Combination in Experimental Cell Models of Human Adrenocortical Cancer. Front Endocrinol (Lausanne). 2021 Apr 26;12:669426. doi: 10.3389/fendo.2021.669426. eCollection 2021. PMID 33981288